CLINICAL TRIAL: NCT01286961
Title: The Interval Between the Time of Second PEG Dose and the Start of the Colonoscopy
Acronym: TOSP
Status: Completed | Type: Observational
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Eun Hee Seo, fellow, Inje University
Other Study IDs: HGI 2011-02
Record Dates: First submitted 2011-01-31; First posted 2011-02-01 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: The Timing of Bowel Preparation in Outpatient Colonoscopy
Keywords: Bowel preparation; Polyethylene glycols; Colonoscopy; Outpatient
MeSH Terms: interventions — Golytely

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- outpatient colonoscopy, bowel preparation, split dose PEG: adult outpatients who undergo colonoscopy
  Interventions: Drug: bowel preparation using split dose of polyethylene glycol

INTERVENTIONS:
Drug: bowel preparation using split dose of polyethylene glycol — polyethylene glycol, split dose(2L/2L), each dose for 1-2hours
  Other Names: Colyte

SUMMARY:
As the duration of the interval between the time of last preparation-agent dose and the start of the colonoscopy is increasing, the quality of bowel preparation will be worse.

DETAILED DESCRIPTION:
The aim of the present studies is to determine how the duration of the interval of the time of last preparation dose and the start of colonoscopy affects the quality of the bowel preparation and when the proper timing of the colonoscopy is after completion of last preparation regimen

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients(18-85 years of age) who undergo colonoscopy for screening, cancer surveillance or with gastrointestinal symptoms, other symptoms

Exclusion Criteria:

* age under 18 years, pregnancy, breast feeding, prior history of surgical large bowel resection, severe renal failure (creatinine ≥ 3.0mg/dL (normal 0.8-1.4)), drug addiction or major psychiatric illness; allergy to PEG, refusal of consent to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult outpatients who undergo colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Quality of bowel preparation according to Ottawa scale | 6 months
  The primary end point of the study was to assess the quality of bowel preparation according to the Ottawa scale, including cleanliness and fluid quantity.

SECONDARY OUTCOMES:
Proper timing of colonoscopy | 6 months
  The secondary end points was to determine the proper interval between the completion of spliting bowel preparation and the start of colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Tae Oh Kim, Ph.D., Study Director — Inje University School of Medicine, Haeundae Paik Hospital, Internal Medicine; Eun Hee Seo, M.D., Principal Investigator — Inje University School of Medicine, Haeundae Paik Hospital, Internal Medicine
Locations (1):
- Haeundae Paik Hospital, Busan, South Korea